CLINICAL TRIAL: NCT05420532
Title: Designing Virtual Reality-based Testing and Rehabilitation for Upper Extremity Software for People With Multiple Sclerosis
Brief Title: Designing Virtual Reality-based Software for People With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuzuncu Yil University (Other)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Asiye Tuba Ozdogar, PhD, Dokuz Eylul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/14-02
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; virtual reality; exergaming
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exergaming Group (Experimental): A video game-based physical activity training will be applied under a physiotherapist supervision for 1 days/week for 8 weeks.
  Interventions: Other: Exergaming

INTERVENTIONS:
Other: Exergaming — A video game-based physical activity training applied using a commercial game console.

SUMMARY:
The study aims to designing virtual reality-based testing and rehabilitation software for people with multiple sclerosis and assess the feasibility of software. Also, the effects of an 8-week virtual reality-based upper extremity training in persons with multiple sclerosis will be investigated.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, inflammatory, and demyelinating disorder that requires long-term rehabilitation. Numerous systematic reviews on MS have demonstrated the effectiveness of rehabilitation strategies such as exercise training, physical therapy, occupational therapy, and multidisciplinary therapy. However, despite the importance of upper extremity performance in daily functional activities, rehabilitation of people with MS (pwMS) generally focuses more on gait and balance, and upper extremity problems remain in the background.

In addition, rehabilitation treatments for pwMS are described as very long and systematic, leading to loss of motivation and adjustment. As a result, technology-based rehabilitation systems such as virtual reality (VR) have been promising in recent years and can provide person-centered task-oriented rehabilitation without needing a device or controller.

In pwMS, physiotherapy and rehabilitation programs based on today's VR studies are usually prepared with game software for computer users without physical disabilities. However, the number of these studies based solely on classical game software has a limited place in treating patients today and is considered insufficient. Moreover, this software is complicated for patients, has a fast-paced structure, and fails to provide disability-focused education or meet patient needs.

For this reason, it is necessary to develop specific game software for pwMS. The study aims to develop virtual reality exergame software for upper extremity rehabilitation in pwMS and evaluate the usability.

Persons who are followed by the outpatient Multiple Sclerosis Clinic of Dokuz Eylül University Hospital will participate in the study. Fifteen participants will be included to determine the feasibility of the software, and they will experience the system for one session. Then 15 participants will be included to investigate the effects of software on upper extremity functions during 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Having a definitive diagnosis of MS according to the 2017 McDonald criteria
* Being over 18 years old
* To be willing to participate in the study.

Exclusion Criteria:

* Having a neurological disease other than MS
* Cognitive disability at a level that hinders assessment and treatment.
* Having a relapse 30 days before or during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Nine-Hole Peg Test | Change from Baseline at 8 weeks
  The Nine-Hole Peg Test is used to assess manual dexterity performance. It requires participants to repeatedly place and then remove nine pegs into nine holes, one at a time, as quickly as possible. Two trials for each hand are performed and the score is the average time. Higher scores indicate less manual dexterity performance.

SECONDARY OUTCOMES:
Jamar Hand Dynamometer | Change from Baseline at 8 weeks
  The Jamar Hand Dynamometer will be used to measure isometric force and peak strength.
Arm Function in Multiple Sclerosis Questionnaire | Change from Baseline at 8 weeks
  Arm Function in Multiple Sclerosis Questionnaire is a unidimensional 31-item questionnaire for measuring arm function in MS. The total sum score ranged from 31 to 186 and a high score indicates a low degree of arm function.
The User Satisfaction Evaluation Questionnaire | immediately after the session
  The User Satisfaction Evaluation Questionnaire, consisting of six questions, will be used to assess the user's satisfaction with the system and exergaming.

OTHER OUTCOMES:
Expanded Disability Status Scale | At baseline
  The Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis. The scale is based on a neurological examination by a clinician. It has steps from 0 to 10. The higher scores indicate higher neurological disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided